CLINICAL TRIAL: NCT01120535
Title: Crux Biomedical Evaluation of the Crux Inferior Vena Cava Filter System 4 (RETRIEVE 4)
Brief Title: Crux Biomedical Evaluation of the Crux Inferior Vena Cava Filter 4
Acronym: RETRIEVE 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crux Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Crux04
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2012-02

CONDITIONS: Pulmonary Embolism
Keywords: Vena Cava; Vena Cava Filter; Pulmonary Embolism; Venous Thromboembolism; Risk of Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism | interventions — Vena Cava Filters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Crux Vena Cava Filter System (Experimental): Subjects at risk for Pulmonary Embolism
  Interventions: Device: Inferior Vena Cava Filter

INTERVENTIONS:
Device: Inferior Vena Cava Filter — Inplant of filter in inferior vena cava.

SUMMARY:
The purpose of this study is to determine if the Crux Vena Cava Filter System is safe and effective in preventing pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a permanent or temporary risk of Pulmonary Embolism.
* Patient must provide informed consent At least one of the following conditions -
* Proven PE
* Recurrent PE despite adequate
* Contraindication to anticoagulation
* Inability to achieve/maintain therapeutic anticoagulation
* Iliocaval DVT
* Large, free-floating proximal DVT
* Massive PE treated with thrombolysis/thrombectomy
* Chronic PE treated with thrombectomy
* Protection during thrombolysis for iliocaval DVT
* PE with limited cardiopulmonary reserve
* Poor compliance with anticoagulation medication
* High risk of injury worsening on anticoagulation
* Multi-trauma patient with high risk of PE
* Surgical patients at high risk of PE
* Medical condition with high risk of PE Patients with a documented vena cava diameter of 17-28mm Patient has IVC anatomy suitable for infra-renal placement Patient is willing to be available for the appropriate follow up

Exclusion Criteria:

* Age <18 years old
* Patient has any one of the following conditions:

  * Renal vein thrombosis
  * IVC thrombosis extending to the renal veins
  * Duplicate IVC
  * Gonadal vein thrombosis
  * Requires supra-renal placement
* Vena cava diameter of 17-28mm
* Uncontrolled infectious disease
* Risk of aseptic PE
* Uncontrolled coagulopathy
* Existing inferior vena cava filter implant
* Life expectancy less than 6 months
* Pregnant or planning a pregnancy in the next 6 months
* Condition that inhibits radiographic visualization of the IVC
* Known allergy or intolerance to polytetrafluoroethylene (PTFE) or Nitinol
* Known hypersensitivity to contract which cannot be pretreated
* Access vessels preclude same insertion of delivery system
* Participation in another drug or device trial
* Unable or unwilling to cooperate with study procedures or required follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 6 Months
  Clinical Success is a composite endpoint consisting of technical success with freedom from pulmonary embolism, filter migration and device related events requiring intervention.

SECONDARY OUTCOMES:
Rates of complications related to vena cava filter use. | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Royal Brisbane Womens Hospital, Brisbane
  - The Alfred Hospital, Melbourne
- Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- See also: Smouse H, Mendes R, Bosiers M et al. The RETRIEVE Trial: Safety and Effectiveness of the Retrieval Crux Vena Cava Filter. JVIR 2013; 24:609-621. — http://www.ncbi.nlm.nih.gov/pubmed/23622035